CLINICAL TRIAL: NCT02671331
Title: The Effect of Loop Duodenal Switch Surgery in Morbidly Obese Patients on Weight Loss at One Year
Brief Title: Loop Duodenal Switch Surgery in Morbidly Obese Patients
Status: Terminated | Type: Observational
Why Stopped: Principal investigator terminated study due to low enrollment.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Tammy Kindel, Assistant Professor, Surgery, Medical College of Wisconsin
Other Study IDs: PRO25874
Record Dates: First submitted 2015-12-29; First posted 2016-02-02 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Type-2 Diabetes Mellitus
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Loop duodenal switch — The loop duodenal switch (L-DS) is a single anastomosis duodeno-intestinal bypass. In this simplified version of a BPD-DS, a sleeve gastrectomy is followed by a single anastomosis of the duodenum to the ileum in a loop fashion. The proposed benefits of this are to reproduce the excellent weight loss seen after a BPD-DS (an accepted and utilized bariatric procedure in the USA) but with the potential for reduced complications. With one anastomoses in the L-DS over two in the BPD-DS there is a theoretical lower probability of leaks, strictures, reduced anesthesia with shorter operative times, and decreased risk of internal hernia.

SUMMARY:
The loop duodenal switch (L-DS) is a single-anastomosis biliopancreatic diversion with duodenal switch (BPD-DS) procedure. The original BPD-DS has two-anastomosis and is an accepted and approved bariatric procedure by the American Society of Metabolic and Bariatric Surgery. Preliminary data from Sanchez-Pernaute et al. (2013) indicates that the L-DS procedure is safer and easier to perform as it only requires one anastomosis compared to the BPD-DS, and offers good results for treatment of both morbid obesity and its metabolic comorbidities, including type-2 diabetes mellitus. However, the initial publications of the loop DS still resulted in a small number of patients with total protein malnutrition. For this reason, the investigators will study the loop DS with a modification of the originally published technique with a longer common channel limb (300 cm) to reduce the risk of protein malnutrition For patients with a BMI >50, many are limited to just a sleeve gastrectomy as other bariatric procedures are technically challenging with increased operative risk. A loop duodenal switch may be a safer operation with improved weight loss for the super-morbidly obese patient.

DETAILED DESCRIPTION:
Screening and Informed Consent

Subjects will be screened on a weekly basis for eligibility of enrollment. If eligible, patients will be approached by study staff at the initial surgical consultation. The purpose of the study and risks of the procedures will be explained to the subject and the consent process must be documented accordingly in the medical record. Subjects who agree to study participation must sign an IRB-approved informed consent form. Subjects will be informed that their participation in this study is voluntary and they may refuse to participate or discontinue from the study at any time. Subjects will be given the opportunity to ask the investigator questions so that they are adequately informed about the research. A copy of the signed informed consent must be provided to the subject and the informed consent process will be documented in source documents. If new information becomes available that may affect a subject's decision to continue to take part in the study, this information will be discussed with the subject by the investigator.

Failure to meet submission requirements:

Each patient will be required to meet their individual insurance companies requirements for submission of bariatric surgery approval. Subjects who provide study consent but then do not submit for insurance approval or are denied will be considered "discontinued" and will not require additional study follow-up visits. The reason for the discontinuation will be clearly delineated on the applicable case report form. Subjects in who the loop duodenal switch procedure is begun but not completed will be considered "discontinued" once discharged from the hospital and not require any additional study follow-up visits. Reasons for discontinuation will be recorded in the case report form.

Additionally, female patients of child bearing age will undergo a standard of care pregnancy test at the time of the pre-operative surgical testing (2/3 weeks before surgery) and always the morning of surgery by urine HCG.

Surgical Procedures:

The operation will be performed per standard of care and as previously described (1-3), with the exception that in this protocol the duodeno-intestinal anastomosis will be performed at approximately 300 cc with moderate stretch from the ileocecal valve, rather than 200 cm or 250 cm, as in previous reports (Cottam et al, 2015). The purpose of this change is to allow greater nutrient absorption since a previous report observed no difference in mean excess weight loss between 200 cm and 250 cm (3). In addition, the sleeve gastrectomy will be performed over a 40 French bougie. The duodeno-intestinal anastomosis will be hand-sewn.

Subjects will be maintained on a low-calorie diet for the first post-operative month, as per standard of care. In addition, multivitamin supplements, calcium, and iron should be prescribed and maintained per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18-70 years of age at time of enrollment.
2. The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent.
3. The subject is under consideration for surgery for obesity or metabolic disease and elects to undergo a primary loop duodenal switch procedure or as a conversion procedure for failed, sustained weight loss after a sleeve gastrectomy or laparoscopic adjustable gastric band performed more than 12 months prior to time of evaluation.
4. The subject has a BMI of greater than or equal to 40 kg/m2 at time of surgical consultation.

Exclusion Criteria:

1. Subjects under 18 years of age or older than 70 years of age.
2. Subject is not willing or able to participate in the study procedures and understand the informed consent.
3. The subject wishes to under a different bariatric procedure other than the loop duodenal switch.
4. The subject has a BMI of less than 40 kg/m2 at the time of surgical consultation.
5. Any female subject who is pregnant, or is actively breast-feeding
6. Any subject who is considered to be part of a vulnerable population (eg. prisoners or those with psychological concerns or those without sufficient mental capacity)
7. The procedure is an emergency procedure
8. The subject is unable to unwilling to comply with the study requirements or follow-up schedule.
9. The subject has comorbidities which, in the opinion of the investigator, will not be appropriate for the study (eg. severe cardiovascular disease or history of gastrointestinal malignancy, history of upper GI gastric surgery, history of intestinal surgery, open cholecystectomy, immunosuppression, and non-ambulatory).
10. The subject has an estimated life expectancy of less than 6 months.
11. The subject has participated in an investigational drug or device research study within 30 days of enrollment.
12. The subject's insurance company does not cover a duodenal switch operation as treatment for morbid obesity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for bariatric surgery and meet inclusion criteria for the Loop duodenal swith surgery with be approached for study consent.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Excess weight loss (EWL) | 12 months post-procedure
  Excess weight loss is a common metric for reporting weight loss after bariatric surgery. The EWL is calculated from an ideal body mass index (BMI) of 25 kg/m^2 and considers weight before surgery and at 12 months post-procedure.

SECONDARY OUTCOMES:
Loop duodenal switch related adverse events | 12 months post-procedure
  Surgery related events such as hospital re-admission, re-operation, complications, etc.
Resolution rate of obesity related co-morbidities | 12 months post-procedure
  Resolution of obesity related co-morbidities including type 2 diabetes mellitus, hypertension, sleep apnea, hyperlipidemia, and other obesity-associated co-morbidities.
SF-36 Quality of Life Survey | 12 months post-procedure
  Quality of life will be measured using the SF-36 Quality of Life Survey.
Gastro-esophageal Reflux Disease Health Related Quality of Life Survey | 12 months post-procedure
  GERD related quality of life will be measured using the Gastro-esophageal Reflux Disease Health Related Quality of Life Survey.
Gastrointestinal Symptoms Rating | 12 months post-procedure
  Gastrointestinal Symptoms will be measured using the Gastrointestinal Symptoms Rating Scale.
Protein malnutrition | 12 months post-procedure
  Protein malnutrition will be assess by albumin level (hypoalbuminemia, <3.5 g/dL) and serum total protein levels (<6.1 g/dL) when oral intake is adequate ( protein intake of 60g +per day).

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Kindel, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Pernaute A, Rubio Herrera MA, Perez-Aguirre E, Garcia Perez JC, Cabrerizo L, Diez Valladares L, Fernandez C, Talavera P, Torres A. Proximal duodenal-ileal end-to-side bypass with sleeve gastrectomy: proposed technique. Obes Surg. 2007 Dec;17(12):1614-8. doi: 10.1007/s11695-007-9287-8. Epub 2007 Nov 27. PMID 18040751
- [Background] Sanchez-Pernaute A, Herrera MA, Perez-Aguirre ME, Talavera P, Cabrerizo L, Matia P, Diez-Valladares L, Barabash A, Martin-Antona E, Garcia-Botella A, Garcia-Almenta EM, Torres A. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S). One to three-year follow-up. Obes Surg. 2010 Dec;20(12):1720-6. doi: 10.1007/s11695-010-0247-3. PMID 20798995
- [Background] Sanchez-Pernaute A, Rubio MA, Perez Aguirre E, Barabash A, Cabrerizo L, Torres A. Single-anastomosis duodenoileal bypass with sleeve gastrectomy: metabolic improvement and weight loss in first 100 patients. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):731-5. doi: 10.1016/j.soard.2012.07.018. Epub 2012 Aug 7. PMID 22963820
- [Background] Cottam A, Cottam D, Medlin W, Richards C, Cottam S, Zaveri H, Surve A. A matched cohort analysis of single anastomosis loop duodenal switch versus Roux-en-Y gastric bypass with 18-month follow-up. Surg Endosc. 2016 Sep;30(9):3958-64. doi: 10.1007/s00464-015-4707-7. Epub 2015 Dec 22. PMID 26694182